CLINICAL TRIAL: NCT04437264
Title: Intermittent Versus Continuous Enteral Nutrition in Mechanically Ventilated Patients in the Medical Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000027328
Record Dates: First submitted 2020-05-19; First posted 2020-06-18 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Enteral Feeding; Nutrition Disorders
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The care team and study staff in the ICU will be aware of arm assignment. Study staff abstracting outcome data will be blinded to arm assignement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent feed (Experimental): Patients will be assigned to receive intermittent enteral feeding protocol. They will receive four equal volume feeds at 8:00, 12:00, 16:00, and 20:00 hours.
  Interventions: Dietary Supplement: Intermittent feed participant
- Continuous feeds (Experimental): Patients will be assigned to receive continuous enteral feeding protocol. Typical goal rates are in the range of 60 to 80 mL per hour for 24 hours per day.
  Interventions: Dietary Supplement: Continuous feeds participant

INTERVENTIONS:
Dietary Supplement: Intermittent feed participant — Patients will be assigned to receive intermittent enteral feeding protocol. They will receive four equal volume feeds at 8:00, 12:00, 16:00, and 20:00 hours.
  Arms: Intermittent feed
Dietary Supplement: Continuous feeds participant — Patients will be assigned to receive continuous enteral feeding protocol. Typical goal rates are in the range of 60 to 80 mL per hour for 24 hours per day.
  Arms: Continuous feeds

SUMMARY:
Evaluate effective delivery of goal nutrition with intermittent as compared with continuous enteral nutrition schedules, as defined by percentage of recommended calories that patient receives per day of interest.

DETAILED DESCRIPTION:
Eligible patients will be approached and if the patient (or surrogate decision maker) is interested, then consent will be obtained for participation in the study. The patient will then be randomly assigned to receive usual care (continuous feeds) or intervention (intermittent feeds, see details below). Randomization will occur via simple block randomization within the REDCap software. Group assignment will not be revealed to the clinical team until the decision to feed the patient has occurred and the actual feeding order is entered. When the clinical team decides to initiate enteral nutrition, they will place a nutrition consult order for tube feed recommendations. Nutrition consult will place recommendations for both continuous feeding and for intermittent schedule, including enteral nutrition formula and dosing. Prior to feeds being started, the patient's randomization status will be revealed to the clinical team. The covering provider will then place the order for enteral nutrition according to the nutritionist's recommendations for the correct feeding schedule.

For patients randomized to continuous feeds, their enteral nutrition will be ordered and delivered as per usual care and standard MICU procedure. Nutritionist will provide recommendations for initiation rate, up titration schedule, and maintenance dosing to be delivered continuously over 24 hours. Under usual care of ICU patients, our clinical nutritionists provide a specified formula, a specified calorie goal, and a suggested titration rate. This is typically 20 mL per hour to start with an increase in rate of 20 mL per hour every 6 to 8 hours until the goal rate is achieved. Typical goal rates are in the range of 60 to 80 mL per hour for 24 hours per day.

For patients randomized to the intervention group (intermittent feeds), they will receive their enteral nutrition according to a research protocol schedule. This will involve the total recommended feed volume divided into four equal volume "meals." These will be delivered at a rate of 400 cc/hr at 8:00, 12:00, 16:00, and 20:00. The up-titration schedule will be as follows: first meal will be 100 mL, and the volume of each meal thereafter will be increased by 100mL until patient is at goal volume (typically between 300 and 450 mL). There are no formula or diets that are inappropriate to be administered on an intermittent feed schedule. The intervention will not change formula selection or total calorie goals. It will only change the schedule of feeding. For all patients, regardless of feeding schedule, the Kangaroo E-Pump will be used to deliver enteral nutrition, and the above rate and volume parameters can be programmed in.

There will be no change in delivery of enteral free water or medications. This schedule will be determined by nursing and clinical care team, as is the current standard of care. To assure correct ordering of intermittent feeds and the insulin prior to each meal, an EPIC orderset with prepopulated instructions will be developed.

If there are no signs of or clinical concerns for intolerance, patients will continue to receive enteral nutrition according to assigned schedule until they are extubated or until enteral nutrition is discontinued.

ELIGIBILITY:
INCLUSION CRITERIA

* MICU Yale New Haven Hospital
* Age >= 18 years old.
* Patients mechanically ventilated via endotracheal tube
* Patients intubated within 72 hours of hospital admission
* First intubation of current hospitalization
* First MICU admission of current hospitalization

EXCLUSION CRITERIA

• Patient has opted out of research participation via institutional patient portal.

At significant risk for gastrointestinal intolerance of intermittent bolus feeds:

* Prior upper gastrointestinal surgery that alters proximal GI anatomy (including but not limited to gastric bypass surgery, gastric banding, complete or partial gastrectomy, Whipple procedure; of note, appendectomy and cholecystectomy are not exclusion criteria.
* Structural gastrointestinal obstruction (such as tumor).
* Chronic enteral nutrition (prior to current admission).
* History of significant esophageal dysmotility (history of GERD is acceptable) or clinically significant GE junction incompetence
* Unable to have head of bed elevated at least 30 degrees while intubated and being fed (this is standard protocol).
* Enteral access terminates post-pyloric (ie nasojejunal or jejunostomy tubes are to be excluded) or unable to place gastric tube for access. (The clinical team will determine type of tube placement. As this is particularly selected by intensivists for patients at higher aspiration risk, this tube enteral access exclusion de facto excludes patients at high aspiration risk.)
* History of small bowel obstruction or ileus on current admission or within last 1 month.
* History of gastroparesis.
* Percutaneous gastrostomy tube or tracheostomy.
* History of ongoing aspiration as determined by a speech medicine specialist or other medical professional or a patent who required adjustment of diet (e.g., thickening of liquids) prior to hospitalization.
* History of significant esophageal dysmotility (history of GERD is acceptable) or clinically significant GE junction incompetence

Other Exclusion Criteria:

* At risk of refeeding syndrome.
* Pregnant patients.
* Patients receiving neuromuscular blockade.
* Patients with glycemic emergency (HHNK, DKA, severe hypoglycemia resulting in MICU admission) or patients controlling their sugar / insulin dosing via continuous glucose monitoring
* Post cardiac arrest (on current admission).
* Received >= 6 hours of enteral nutrition (regardless of volume) at the time of screening and team is able to consent / enroll / initiate intermittent feed within an additional 2 hours.
* Plan for extubation within 24 hours.
* Not English-speaking.
* Patients otherwise excluded by the treating physician.
* Retrospective exclusion: patients who initially met eligibility criteria, but no nutrition consult (i.e., decision to initiate feeds by clinical providers) placed within 72 hours of intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Recommended calories | Intubation day 1 to intubation day 10
  percentage of recommended calories that patient receives per day of interest during study period

SECONDARY OUTCOMES:
Percentage of patients with aspiration | Intubation day 1 to intubation day 10
  percentage of patients experiencing aspiration
Percentage of patients experiencing intolerance of feeding | Intubation day 1 to intubation day 10
  percentage of patients experiencing intolerance of feeding including nausea, vomiting, diarrhea, ileus
feasibility: proportion complete protocol | Intubation day 1 to intubation day 10
  percentage of patients assigned to intervention (ie intermittent feeding protocol) that remain on study protocol for study period of interest.
delirium | intubation day 1 until 14 days later
  number of delirium and coma free days out of 14 following intubation
urine 6-sulfatoxymelatonin acrophase | day 1 to 3 following initiation of feeds
  Urine 6-sulfatoxymelatonin acrophase defined as the time of fitted peak 6-sulfatoxymelatonin from fitting a cosine curve to hourly urine aMT6s levels will be determined daily
maximum glucose | Intubation day 1 to intubation day 10
  highest glucose per day of interest
minimum glucose | Intubation day 1 to intubation day 10
  lowest glucose per day of interest
insulin usage | Intubation day 1 to intubation day 10
  number of insulin units used per day (composite of short and long acting formulations)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P Knauert, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, York Street Campus, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data can be made available upon request.